CLINICAL TRIAL: NCT05875662
Title: Evaluation of Pulmonary Ventilation After Fiberoptic Bronchoscopy in Critically Ill Patients Using Electrical Impedance Tomography
Brief Title: Pulmonary Ventilation After Fiberoptic Bronchoscopy Using EIT
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Shan Lv, Principal Investigator, Peking University People's Hospital
Other Study IDs: PekingUPH-2023z038
Record Dates: First submitted 2023-05-07; First posted 2023-05-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Bronchoscopy; Atelectasis; Mechanical Ventilation
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanical ventilation patients undergoing fiberoptic bronchoscopy: After being included in the patient, the EIT chest strap was worn to measure the end expiratory lung impedance and tidal impedance variable, assess the distribution of lung ventilation in patients and record GI index and CoV. EELI,TIV, GI index, CoV, vital signs of patients, including heart rate, blood pressure, respiratory rate, SpO2, ventilator parameters, including mode, driving pressure, FiO2, PEEP, and lung compliance was recorded before and after bronchoscopy. Patients underwent a recruitment maneuver 5 minutes after bronchoscopy maintaining breaths at a PC of 40 cm H2O with PEEP of 20 cm H2O in pressure control mode for 1 minute, then, PEEP was decreased from 20 to preceding PEEP value in steps of 2 cm H2O with a duration of at least 10 breaths or 30 seconds at each step.

SUMMARY:
Background: Fiber bronchoscopy is a routine operation in intensive care unit (ICU), but it may cause local collapse of the lung. Recruitment maneuver (RM) after fiber bronchoscopy may have the potential to restore functional residual air volume and increase lung volume. However, there is still a lack of quantitative indicators to evaluate the effect of recruitment maneuver. With electrical impedance tomography (EIT), we can monitor lung ventilation in real time to understand the situation of lung ventilation.

Objective: To evaluate whether recruitment maneuver after fiber bronchoscopy can improve lung volume and improve lung ventilation, and which people are most likely to benefit from it, by monitoring the end expiratory pulmonary impedance of critically ill patients undergoing bedside fiber bronchoscopy to monitor the lung ventilation before and after the operation and before and after recruitment maneuver.

Study Design: A prospective observational study was conducted to monitor the end expiratory lung impedance (EELI), tidal impedance variable (TIV), global inhomogeneity (GI) index and Center of Ventilation (CoV) before and after bronchoscopy and recruitment maneuver, and then to understand the changes of lung volume and ventilation.

DETAILED DESCRIPTION:
At present, people pay more and more attention to the atelectasis caused by the sputum suction operation of fiberoptic bronchoscope. A recent observational study confirmed that more than 80% of patients will have atelectasis in at least one lung segment after the completion of the bronchoscope operation using the imaging method of cluster computed tomography (CT). The production of atelectasis will affect the patient's subsequent ventilation function, causing hypoxemia. Pulmonary atelectasis is a commonly used procedure for patients with acute respiratory distress syndrome (ARDS) to restore lung volume and improve atelectasis. Therefore, it is worth exploring whether adopting recruitment maneuver after bronchoscopy can avoid or reduce the problems of subsequent lung collapse and atelectasis in patients, and how to quantify it.

electrical impedance tomography, referred to as EIT, is a new imaging technology that can be implemented at the bedside in real-time, non-invasive and radiation free. The basic principle is to apply a weak current through local electrodes to sense the changes in the chest bioelectrical impedance during breathing, and then use the corresponding imaging algorithm to monitor the status of ventilation function in different areas of the lung, which is presented in real-time dynamic lung tomography ventilation images. Previous studies have found that through EIT, the end expiratory lung impedance (EELI) of the lungs can be monitored, indirectly reflecting the end expiratory volume of the lungs, thereby achieving the goal of monitoring local lung collapse caused by fiberoptic bronchoscope.

After being included in the patient, the EIT chest strap was worn to measure the end expiratory lung impedance and tidal impedance variable before bronchoscopy, and recorded as EELI before and TIV before, global inhomogeneity (GI) index ,Center of Ventilation (CoV), the vital signs of patients, including heart rate, blood pressure, respiratory rate, SpO2, ventilator parameters, including mode, PC/Vt, FiO2, PEEP, and lung compliance before bronchoscopy were recorded. Prepare fiber bronchoscopy and perform fiber bronchoscopy according to routine procedures in ICU. Record the duration of fiberoptic bronchoscopy examination and the condition of secretions.

After the fiber bronchoscopy examination, the end expiratory lung impedance and tidal impedance variables were recorded as EELI after operation and TIV after operation. The GI index, CoV, vital signs of patients, including heart rate, blood pressure, respiratory rate, SpO2, ventilator parameters, including mode, PC/Vt, FiO2, PEEP, and compliance were recorded. Perform recruitment maneuver using PCV mode, PEEP 20 cmH2O, PC 20 cmH2O, for 1 minute, then gradually reduce the ventilator pressure and restore the mode and parameters before bronchoscopy. If complications occur during the process of recruitment maneuver, timely record them. End expiratory lung impedance and tidal impedance variables were recorded as EELI after recruitment and TIV after recruitment. The GI index, CoV, vital signs of patients, including heart rate, blood pressure, respiratory rate, SpO2, ventilator parameters, including mode, PC/Vt, FiO2, PEEP, and compliance were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive mechanical ventilation undergoing fiberoptic bronchoscopy in ICU

Exclusion Criteria:

* Age<18 years old or>85 years old
* Pregnant women
* Patients undergoing emergency bronchoscopy examination
* Patients who undergo bronchoscopy only to confirm the position of the artificial airway
* Patients who are unable to wear EIT chest straps due to surgical incisions or closed drainage tubes in the chest
* Patients who refuse to participate in this trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasive mechanical ventilation patients admitted to the ICU who plan to undergo bedside fiberoptic bronchoscopy
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The change in end-expiratory lung impedance (ΔEELI) | Changes in EELI within 5 minutes before and 5 minutes after lung recruitment maneuver
  EIT was performed with a PulmoVista 500(Drager Medical, Lübeck, Germany).The signals were recorded and later reviewed offline using a dedicated software program (Dräger Medical GmbH EIT data analysis version 6.3).ΔEELI refers to differences in end-expiration lung impedance between 5 minutes before and 5 minutes after lung recruitment maneuver.
The change in tidal impedance variable (ΔTIV) | Changes in TIV within 5 minutes before and 5 minutes after lung recruitment maneuver
  TIV, which correlates with gas volume changes in the lung, was calculated by selecting 10 subsequent breathing cycles from the recorded EIT sequences. Thereafter, differences in global impedance between end-inspiration and end-expiration were calculated, then averaged.ΔTIV is the change in TIV within 5 minutes before and 5 minutes after lung recruitment maneuver

CONTACTS AND LOCATIONS:
Overall Officials: Shan Lyu, Master, Principal Investigator — Peking University People's Hospital
Locations (1):
- Department of Critical Care Medicine, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No